CLINICAL TRIAL: NCT00224640
Title: Effect of Iron-Chelating Therapy in Friedreich Ataxia. Study Phase I/II
Brief Title: Iron-Chelating Therapy and Friedreich Ataxia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel Ouslimany, Department Clinical Research of Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P041201; PCR 05001
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2007-03

CONDITIONS: Friedreich Ataxia
Keywords: Iron-chelating treatment
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Iron chelating intervention
  Interventions: Drug: Iron chelating intervention

INTERVENTIONS:
Drug: Iron chelating intervention — Iron chelating intervention

SUMMARY:
Friedreich ataxia, an autosomal recessive condition, ascribed to frataxin gene expansion, has been shown to result from an iron- induced injury to the mitochondrial respiratory chain. Buffering free radicals with short-chain quinones (Idebenone) protects the patients against cardiomyopathy but not CNS involvement. Removing CNS iron should limit the impact of the neurological symptoms of the disease.

DETAILED DESCRIPTION:
The current clinical trial is a monocentric open phase1-2 trial in the context of rare diseases framework, aimed to the goal of defining the tolerance/efficacy of the treatment.

Inclusion criteria: minimum age: 13 years Follow up in the Dept of Genetics, Hospital Necker-Enfants Malades, Paris, France

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age: 13 years
2. Molecular confirmation of frataxin gene mutation
3. Iron overload evaluation
4. Presence of lactate
5. Echography response to Idebenone treatment
6. Urinary test of pregnancy for girls
7. Sexual abstinence for men
8. Information consent

Exclusion Criteria:

1. No disturbance of iron metabolism
2. No response to Idebenone
3. Friedreich not confirmed
4. Polynuclear neutrophils <2 x 109/L or hemoglobin < 8g/dL
5. No participation to other trial
6. Doubt regarding the compliance of the patient to protocol
7. Impossibility to undergo X-ray examination or presence of iron material in the backbone
8. Pregnant women
9. Absence of social insurance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
assessment of iron overload at TO and month2 by imagery | at months :0, 1 ,2 ,4 ,6

SECONDARY OUTCOMES:
Clinical (monthly) and biological parameter follow- up ( blood count, | weekly
plasma iron, ferritin, transferrin and liver enzymes) | every months

CONTACTS AND LOCATIONS:
Overall Officials: Arnold MUNNICH, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, France